CLINICAL TRIAL: NCT06132685
Title: Post-Operative Dosing of Steroids Post Craniotomy for Brain Tumor (PODS)
Brief Title: Post-Operative Dosing of Dexamethasone in Patients With Brain Tumors After a Craniotomy, PODS Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kimberly Bojanowski Hoang, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003975; NCI-2023-04702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00003975 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5678-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2023-09-06; First posted 2023-11-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Low Grade Glioma; Malignant Brain Glioma; Malignant Brain Neoplasm; Meningioma
MeSH Terms: conditions — Brain Neoplasms; Meningioma | interventions — Specimen Handling; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (NDS) (Experimental): Patients receive tapering doses of dexamethasone on days 1-15. Patients also undergo blood sample collection at time of surgery, at follow up visits and optionally at wound check visit 10-14 days post operative at investigator availability. Patients additionally undergo MRI and CT scan during inpatient stay as part of standard of care.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dexamethasone; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Arm II (RDS) (Experimental): Patients receive tapering doses of dexamethasone on days 1-4. Patients may receive dexamethasone IV and restart the taper if clinically indicated. Patients also undergo blood sample collection at time of surgery, follow up visits and optionally at wound check visit 10-14 days post operative at investigator availability. Patients additionally undergo MRI and CT scan during inpatient stay as part of standard of care.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dexamethasone; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Dexamethasone — Given dexamethasone or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests the effect of decreasing (tapering) doses of dexamethasone on steroid side effects in patients after surgery to remove (craniotomy) a brain tumor. Steroids are the gold standard post-surgery treatment to reduce swelling (edema) at the surgical site to reduce neurological symptoms. Although, corticosteroids reduce edema, they have side effects including high blood sugar, high blood pressure, and can impair wound healing. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response. It also works to treat other conditions by reducing swelling and redness. Tapering doses dexamethasone may decrease steroid side effects without increasing the risk of edema in patients with brain tumors after a craniotomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to evaluate the efficacy of a reduced dosage steroid schedule (RDS) in patients who have undergone craniotomy for high grade glioma (HGG), low grade glioma (LGG), brain metastasis (BM), and meningiomas as compared with the normal dosing schedule (NDS).

II. RDS after undergoing craniotomy for brain tumor has no impact on length of stay, 30 day readmission, and need for repeat imaging when compared to NDS.

SECONDARY OBJECTIVE:

I. RDS after craniotomy for brain tumor has no impact on development of steroid related side effects (new onset or worsening hypertension, hyperglycemia, wound infection, impaired wound healing, steroid dependence, neuropsychiatric disturbance) when compared to NDS.

TERTIARY/EXPLORATORY OBJECTIVE:

I. RDS after craniotomy has no effect on lymphocyte count and differential at 10-14 days after surgery.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (NDS): Patients receive tapering doses of dexamethasone on days 1-15. Patients also undergo blood sample collection at time of surgery, at follow up visits and optionally at wound check visit 10-14 days post operative at investigator availability. Patients additionally undergo magnetic resonance imaging (MRI) and computed tomography (CT) scan during inpatient stay as part of standard of care.

ARM II (RDS): Patients receive tapering doses of dexamethasone on days 1-4. Patients may receive dexamethasone intravenously (IV) and restart the taper if clinically indicated. Patients also undergo blood sample collection at time of surgery, follow up visits and optionally at wound check visit 10-14 days post operative at investigator availability. Patients additionally undergo MRI and CT scan during inpatient stay as part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiographic findings consistent with either HGG, LGG, Meningioma, or brain metastasis
* Age equal to or above 18

Exclusion Criteria:

* Known hypothalamic-pituitary-adrenal (HPA) axis dysfunction
* Tumor causing compression of the sella or pituitary dysfunction
* Known immunodeficiency - including but not limited to severe combined immunodeficiency (SCID), common variable immunodeficiency (CVID), lymphocytopenia
* Taking immunosuppressive drugs - including but not limited to methotrexate, mycophenolate, rapamycin, tacrolimus, adalimumab, infliximab. Greater than two weeks of recent daily corticosteroid use or the use of corticosteroids equivalent to > 85 mg of dexamethasone in the last month
* Current lymphoma or leukemia
* History of solid organ transplant
* Minors < 18
* Pregnant women
* History of cerebrovascular accident leading to neurologic deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 3 months
  The two-sample t-test or Mann-Whitney U test utilized to estimate the differences between the two groups. General linear model employed in the multivariable analysis to estimate the adjusted difference in length of hospital stay between the two groups after adjusting for other factors.
30-day repeat admission rate | At 30 days after surgery
  Comparison between the two groups assessed using Fisher exact test or Chi-Square test. Logistic regression used to compare between the two groups after adjusting for other factors. Odds ratios (OR) and 95% confidence intervals (CIs) calculated to evaluate the strength of any association.
Need for repeat head imaging | Up to 3 months
  Comparison between the two groups assessed using Fisher exact test or Chi-Square test. Logistic regression used to compare between the two groups after adjusting for other factors. OR and 95% CIs calculated to evaluate the strength of any association.

SECONDARY OUTCOMES:
Incidence of new neurologic deficit | At less than 30 days and at 3 months
  Comparison between the two groups assessed using Fisher exact test or Chi-Square test. Logistic regression used to compare between the two groups after adjusting for other factors. OR and 95% CIs calculated to evaluate the strength of any association.
Breakthrough seizures | Up to 30 days after surgery
  Comparison between the two groups assessed using Fisher exact test or Chi-Square test. Logistic regression used to compare between the two groups after adjusting for other factors. OR and 95% CIs calculated to evaluate the strength of any association.
Evidence of Worsening Cerebral Edema | Between 5 and 30 days after surgery
  This measure will be a three-level scale determined by the final neuroradiology read of comparison imaging as either improved cerebral edema, stable cerebral edema, or worsened cerebral edema when evaluated on repeat CT Head without contrast.
Evaluation for Steroid Dependence | At long term follow up to 3 months after surgery
  This measure will be evaluated in a binary manner as either the patient having been successfully weaned off of all steroids or the patient remaining on supplemental daily steroids due to the inability to wean off of steroids due to symptomatic adrenal insufficiency. The assessment of adrenal insufficiency will not be done as part of this the study, this study will document the continued use of supplemental daily steroids at 3 month follow-up versus not.
Rate of new onset hypertension | During inpatient stay up to 3 months after surgery
  Defined as sustained systolic blood pressure > 140. Comparison between the two groups assessed using Fisher exact test or Chi-Square test. Logistic regression used to compare between the two groups after adjusting for other factors. OR and 95% CIs calculated to evaluate the strength of any association.
Rate of new onset hyperglycemia | During inpatient stay up to 3 months after surgery
  Defined as random blood glucose > 100 and/or new insulin requirement. Comparison between the two groups assessed using Fisher exact test or Chi-Square test. Logistic regression used to compare between the two groups after adjusting for other factors. OR and 95% CIs calculated to evaluate the strength of any association.
Evaluation for Wound infection or Delayed Wound Healing | At 2 week wound check after surgery
  This criterion will be assessed via the "Wound Check Form" which uses a scale from 1-9 with worsening wound healing and infection indicated by an increased score. Modifiers A and B indicating cellulitis and purulence respectively are also added to the scale. The worst score on this scale would therefore be a 9AB, and a perfectly healed wound would be score of 1.
Evaluation for Need for Psychiatric Consult or Neuropsychiatric Side Effects | At 2 week follow up after surgery
  This criterion will be initially assessed via EPIC documentation via daily assessment via Neurosurgery residents whether the patient has experienced severe new onset behavioral issues in the post-op period typically associated with steroids (agitation, psychosis, mania). This will be then categorized into a binary system determining either the presence or absence of new severe agitation, psychosis, or mania. In addition, at the post operative visit, the patient will fill out the 'Dexamethasone Symptom questionnaire' which is a standardized questionnaire recording binary presence vs no presence of a list of common subjective symptoms experienced by patients on chronic steroids (headache, changes in body habitus etc) which will additionally be recorded.
Change in lymphocyte count and differential | At baseline and 10-14 days post-operative
  Compared using the two-sample t-test. A general linear model will be used in the multivariable analysis to estimate the adjusted difference.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hoang, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States